CLINICAL TRIAL: NCT03058029
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effect of Gelesis200 on Body Weight in Overweight and Obese Subjects Without or With Type 2 Diabetes
Brief Title: Effect of Gelesis200 on Body Weight in Overweight and Obese Subjects w/o Type 2 Diabetes
Acronym: LIGHT-UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gelesis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-200-002
Record Dates: First submitted 2017-01-13; First posted 2017-02-20 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Overweight; Diabetes; PreDiabetes; Obesity
MeSH Terms: conditions — Overweight; Diabetes Mellitus; Prediabetic State; Obesity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Gelesis200 (Experimental): Gelesis200: Three (3) Gelesis200 capsules (2.10 gram (g)) two (2) times per day (id est (i.e.), lunch and dinner)
  Interventions: Device: Gelesis200
- Placebo (Placebo Comparator): Placebo: Three (3) placebo capsules two (2) times per day (i.e., lunch and dinner)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Gelesis200 — Subject would take Gelesis200 capsules 2 times per day.
  Arms: Gelesis200
Device: Placebo — Subject would take placebo capsules 2 times per day.
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Assessing the Effect of Gelesis200 on Body Weight in Overweight and Obese Subjects without or with Type 2 Diabetes

DETAILED DESCRIPTION:
Multicenter, two-cohort, randomized, double-blind, placebo-controlled, parallel-group, fixed-dose, adaptive (Two Phases).

In the first Phase of the adaptive design, unblinded interim analyses were conducted on 57 subjects and used to adjust the design for the second Phase. The first Phase was completed under protocol Version 1.0. Data used in the unblinded interim analyses of the first Phase will not be included in the second Phase (protocol Version 2.0 and subsequent protocol versions) analyses.

The study will evaluate the safety, tolerability and efficacy of Gelesis200 as a superabsorbent hydrogel for weight loss in treated diabetic subjects, untreated diabetic subjects, and prediabetic subjects (Cohort 1).

The study will evaluate separately the safety, tolerability and efficacy of Gelesis200 for weight loss in normoglycemic subjects (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Age ≥22 years and ≤65 years
3. Ambulatory
4. BMI ≥27 kg/M2 and ≤40 kg/M2
5. Non-diabetic subjects, including:

   1. Normoglycemic subjects with FPG <100 mg/dL [<5.6 mmol/L] at both Screening Visits with HbA1c <5.7% (<39 mmol/mol), or
   2. Prediabetic subjects with FPG ≥100 mg/dL and <126 mg/dL (≥5.6 mmol/L and ≤7.0 mmol/L) at both Screening Visits with HbA1c ≤6.4% (≤46 mmol/mol) [if only one (1) value is within this range, the other value should not be ≥126 mg/dL (≥7.0 mmol/L) and HbA1c should be ≥5.7% (≥39 mmol/mol) and ≤6.4% (≤46 mmol/mol)]; or Diabetic subjects, including:

   <!-- -->

   1. Untreated subjects with FPG ≤200 mg/dL (≤11.2 mmol/L) at both Screening Visits and either FPG ≥126 mg/dL (≥7.0 mmol/L) at both Screening Visits or FPG <126 mg/dL (<7.0 mmol/L) at one (1) or both Screening Visits with HbA1c ≥6.5% (≥48 mmol/mol), or
   2. Drug-treated subjects with metformin and/or DPP-4 inhibitors with FPG ≥70 mg/dL and ≤270 mg/dL (≥3.9 mmol/L and ≤15.1 mmol/L) at both Screening Visits
6. Ability to follow verbal and written instructions
7. Consent obtained via signed ICF

Exclusion Criteria:

1. Pregnancy (or positive serum or urine pregnancy test(s) in females of childbearing potential)
2. Absence of medically approved contraception in females of childbearing potential (e.g., hysterectomy, oral contraceptive medications, intrauterine device combined with a barrier method, two (2) combined barrier methods such as diaphragm and condom or spermicide, or condom and spermicide; bilateral tubal ligation and vasectomy are acceptable contraceptive methods when combined with a single method above)
3. History of allergic reaction to CMC, citric acid, sodium stearyl fumarate, maltodextrin, gelatin, or titanium dioxide
4. Participation in a weight loss study within the past six (6) months
5. Administration of GSP2, GSP3, Gelesis100, or Gelesis200 in a previous study
6. Administration of investigational products within one (1) month prior to Screening Visit 1
7. Blood transfusion within three (3) months prior to Screening Visit 1
8. Smoking cessation within six (6) months prior to Screening Visit 1 or considering smoking cessation during the study
9. Anticipated surgical intervention during the study period
10. Known Type 1 Diabetes
11. History of eating disorders including binge eating (except mild binge eating) or emesis ≥2/week from any cause within six (6) months prior to Screening Visit 1
12. Weight change ≥3% within three (3) months prior to and during the Screening period
13. Supine SBP >160 mm Hg and/or supine DBP >95 mm Hg
14. Angina, coronary bypass, or myocardial infarction within six (6) months prior to Screening Visit 1
15. History of swallowing disorders within six (6) months prior to Screening Visit 1
16. Esophageal anatomic abnormalities (e.g., webs, diverticuli, rings)
17. History of gastric or duodenal ulcer within six (6) months prior to Screening Visit 1
18. History of gastroparesis (e.g., chronic nausea, vomiting ≥2 occurrences per week, heartburn, etc.) within six (6) months prior to Screening Visit 1
19. History of gastric bypass or any other gastric surgery
20. History of inflammatory bowel diseases
21. History of intestinal stricture (e.g., Crohn's disease)
22. History of intestinal obstruction or high risk of intestinal obstruction, including suspected small bowel adhesions
23. History of pancreatitis within six (6) months prior to Screening Visit 1
24. History of malabsorption within six (6) months prior to Screening Visit 1
25. Laxative users, except those on stable doses within one (1) month prior to Screening Visit 1
26. History of hepatitis B or C within six (6) months prior to Screening Visit 1
27. History of HIV
28. History of cancer within the past five (5) years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer)
29. Any other clinically significant disease interfering with the assessments of Gelesis200 (e.g., disease requiring corrective treatment, potentially leading to study discontinuation)
30. Abnormal serum TSH
31. HbA1c >8.5% (>69 mmol/mol)
32. Serum LDL cholesterol ≥160 mg/dL (≥4.15 mmol/L)
33. Serum triglycerides ≥350 mg/dL (≥3.96 mmol/L)
34. Positive test for drugs of abuse in the urine
35. Any relevant biochemical abnormality interfering with the assessments of Gelesis200
36. Anti-obesity medications (including herbal preparations) within one (1) month prior to Screening Visit 1
37. Systemic corticosteroids within one (1) month prior to Screening Visit 1
38. Thyroid hormones or preparations within one (1) month prior to Screening Visit 1 [except stable dose of replacement therapy for at least two (2) months]
39. TSH suppression therapy for thyroid cancer
40. Estrogen within one (1) month prior to Screening Visit 1 [except stable dose of replacement therapy or contraceptives for at least one (1) month]
41. Any other medication known to cause weight loss or weight gain within one (1) month prior to Screening Visit 1
42. Antidiabetic medications within one (1) month prior to Screening Visit 1 [except stable doses of metformin and DPP-4 inhibitors for at least one (1) month in subjects with Type 2 Diabetes]
43. Change in medications treating hypertension within one (1) month [one (1) week for diuretics] prior to Screening Visit 1
44. Change in medications treating dyslipidemia within one (1) month prior to Screening Visit 1
45. Anticipated requirement for use of prohibited concomitant medications
46. Any other condition that, in the opinion of the Investigator or Sponsor, would interfere with the subject's ability to participate in the study

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with weight loss ≥5.0% | Change from baseline to day 171 (week 25)
  In treated diabetic subjects, untreated diabetic subjects, and pre-diabetic subjects (Cohort 1)
Percent change in body weight | Change from baseline to day 171 (week 25)
  In treated diabetic subjects, untreated diabetic subjects, and pre-diabetic subjects (Cohort 1)

SECONDARY OUTCOMES:
Proportion of subjects with weight loss ≥10.0% | Up to 25 weeks
  In treated diabetic subjects, untreated diabetic subjects, and pre-diabetic subjects (Cohort 1)
Proportion of subjects with weight loss ≥10.0% | Up to 25 weeks
  Treated diabetics (subgroup of Cohort 1)
Proportion of subjects with weight loss ≥10.0% | Up to 25 weeks
  Pre-diabetics and untreated diabetics (subgroup of Cohort 1)
Proportion of subjects with weight loss ≥5.0% | Up to 25 weeks
  Treated diabetic subjects (subgroup of Cohort 1)
Proportion of subjects with weight loss ≥5.0% | Up to 25 weeks
  Pre-diabetics and untreated diabetics (subgroup of Cohort 1)
Percent change in FSI | Up to 25 weeks
  Pre-diabetics and untreated diabetics (subgroup of Cohort 1)
Percent change in insulin AUC during OGTT | Up to 25 weeks
  Pre-diabetic subjects (subgroup of Cohort 1)
Change in HbA1c | Up to 25 weeks
  Diabetic subjects with HbA1c ≥7.5% (≥58 mmol/mol) at baseline (subgroup of Cohort 1)

OTHER OUTCOMES:
Proportion of subjects with weight loss ≥7.5% | Change from baseline to day 171 (week 25)
  In treated diabetic subjects, untreated diabetic subjects, and pre-diabetic subjects (Cohort 1)
Proportion of subjects with weight loss ≥7.5% | Change from baseline to day 171 (week 25)
  In treated diabetic subjects (subgroup of Cohort 1)
Proportion of subjects with weight loss ≥7.5% | Change from baseline to day 171 (week 25)
  Pre-diabetics and untreated diabetics (subgroup of Cohort 1)
Percent change in body weight | Change from baseline to day 171 (week 25)
  In treated diabetic subjects (subgroup of Cohort 1)
Percent change in body weight | Change from baseline to day 171 (week 25)
  Pre-diabetics and untreated diabetics (subgroup of Cohort 1)
Change in waist circumference | Change from baseline to day 171 (week 25)
  In treated diabetic subjects, untreated diabetic subjects, and pre-diabetic subjects (Cohort 1)
Percent change in estimated excess body weight | Change from baseline to day 171 (week 25)
  In treated diabetic subjects, untreated diabetic subjects, and pre-diabetic subjects (Cohort 1)
Change in BMI | Change from baseline to day 171 (week 25)
  In treated diabetic subjects, untreated diabetic subjects, and pre-diabetic subjects (Cohort 1)
Percent change in FSI | Change from baseline to day 171 (week 25)
  In subjects FSI ≥10 µU/mL in both screening visits (subgroup of Cohort 1)
Percent change in HOMA-IR and log HOMA-IR | Change from baseline to day 171 (week 25)
  Pre-diabetics and untreated diabetics (subgroup of Cohort 1)
Percent change in QUICKI | Change from baseline to day 171 (week 25)
  Pre-diabetics and untreated diabetics (subgroup of Cohort 1)
Percent change in fasting serum lipids | Change from baseline to day 171 (week 25)
  Subjects with dyslipidemia defined as LDL ≥130 mg/dL (≥3.37 mmol/L) and/or triglycerides ≥150 mg/dL (≥1.69 mmol/L)] at baseline (subgroup of Cohort 1)
Change in blood pressure | Change from baseline to day 171 (week 25)
  Subjects with hypertension defined as SBP ≥140 mm Hg and/or DBP ≥90 mm Hg) at baseline (subgroup of Cohort 1)
Proportion of subjects with weight loss ≥5.0% | Change from baseline to day 171 (week 25)
  Normoglycemic subjects (Cohort 2)
Percent change in body weight | Change from baseline to day 171 (week 25)
  Normoglycemic subjects (Cohort 2)
Percent change in FSI | Change from baseline to day 171 (week 25)
  Subjects with FSI ≥10 µU/mL at both Screening Visits (subgroup of Cohort 2)
Percent change in insulin AUC during OGTT | Change from baseline to day 171 (week 25)
  Subjects with FSI ≥10 µU/mL at both Screening Visits (subgroup of Cohort 2)
Proportion of subjects with weight loss ≥7.5% | Change from baseline to day 171 (week 25)
  Normoglycemic subjects (Cohort 2)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (12):
  - Central Alabama Research, Birmingham, Alabama
  - Meridien Research, Inc - Bradenton, Bradenton, Florida
  - Baptist Diabetes Associates, P.A., Miami, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - The Center for Pharmaceutical Research, Kansas City, Kansas
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Radiant Research, Cincinnati, Ohio
  - Mountain View Clinical Research - Greer, Greer, South Carolina
  - Volunteer Research Group and New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee
  - SAMCRC, San Antonio, Texas
  - Tarheel Clinical Research, LLC, Sugar Land, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Canada (2):
  - University of Ottawa - Institut de Recherche de l'Hospital d'Ottawa (IRHO) (Ottawa Hospital Research Institute (OHRI)), Ottawa, Ontario
  - Université Laval, Québec, Quebec
- Health&Care, s.r.o, Prague, Czechia
- University of Copenhagen - Department of Nutrition, Exercise and Sports, Frederiksberg, Denmark
- Hungary (3):
  - Qualiclinic Kft, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
- IRCCS Policlinico San Donato, San Donato Milanese, Italy
- Poland (5):
  - NZOZ Specjalistyczny Osrodek Internistyczno - Diabetologiczny, Bialystok
  - NZOZ All - Med Centrum Medyczne Specjalistyczne Gabinety Lekarskie Marcin Ogorek, Lodz
  - MEDICOME Sp. z o.o., Oświęcim
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Centrum Badawcze Wspolczesnej Terapii, Warsaw
- United Kingdom (5):
  - Oakenhurst Medical Practice, Blackburn
  - Ashgate Medical Practice (Research Office), Chesterfield
  - Aintree University Hospital, Liverpool
  - The James Cook University Hospital, Middlesbrough
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: No